CLINICAL TRIAL: NCT01358721
Title: An Exploratory Study to Investigate the Immunomodulatory Activity of Various Dose Levels of Anti Programmed-Death-1 (PD-1) Antibody (BMS-936558) in Subjects With Metastatic Clear Cell Renal Cell Carcinoma (RCC).
Brief Title: Phase I Biomarker Study (BMS-936558)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Collaborators: Ono Pharma USA Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: CA209-009; 2011-005379-18 (EudraCT Number)
Record Dates: First submitted 2011-05-20; First posted 2011-05-24 (Estimated); Results first posted 2019-07-26 (Actual); Last update posted 2021-10-28 (Actual); Status verified 2021-10

CONDITIONS: Renal Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Arm 1: BMS-936558 (Experimental)
  Interventions: Drug: BMS-936558 (Anti-PD-1)
- Arm 2: BMS-936558 (Experimental)
  Interventions: Drug: BMS-936558 (Anti-PD-1)
- Arm 3: BMS-936558 (Experimental)
  Interventions: Drug: BMS-936558 (Anti-PD-1)
- Arm 4: BMS-936558 (Experimental): (treatment naive)
  Interventions: Drug: BMS-936558 (Anti-PD-1)

INTERVENTIONS:
Drug: BMS-936558 (Anti-PD-1) — Solution, Intravenous infusion, 0.3 mg/kg, Every 3 weeks, Indefinitely depending on response
  Arms: Arm 1: BMS-936558
Drug: BMS-936558 (Anti-PD-1) — Solution, Intravenous infusion, 2 mg/kg, Every 3 weeks, Indefinitely depending on response
  Arms: Arm 2: BMS-936558
Drug: BMS-936558 (Anti-PD-1) — Solution, Intravenous infusion, 10 mg/kg, Every 3 weeks, Indefinitely depending on response
  Arms: Arm 3: BMS-936558; Arm 4: BMS-936558

SUMMARY:
The purpose of this study is to evaluate the pharmacodynamic and biologic properties of BMS-936558 in subjects with metastatic renal cell carcinoma.

DETAILED DESCRIPTION:
Intervention Model: Parallel Dose Comparison

ELIGIBILITY:
For more information regarding BMS clinical trial participation, please visit www.BMSStudyConnect.com

Inclusion Criteria:

* Women and men ≥ 18 years of age.
* Histologic confirmation of renal cell carcinoma with a clear cell component.
* Measurable disease as defined by Response Evaluation Criteria in Solid Tumors (RECIST).
* Tumor sites that can be accessed for repeat biopsies at acceptable clinical risk.
* Previously treated subjects must have failed at least 1 prior anti-angiogenic agent and can have a maximum of 3 prior systemic treatments for renal cell cancer.
* Subjects in the treatment naive arm cannot have received prior systemic therapy for their renal cell carcinoma.

Exclusion Criteria:

* Active or progressing brain metastases.
* Active concomitant.
* Active or history of autoimmune disease.
* Active use of systemic corticosteroids.
* Prior therapy with Cytotoxic T lymphocyte-associated antigen 4 (anti-CTLA4), anti Programmed death-1 (anti-PD1), anti Programmed death ligand 1 (anti-PD-L1), anti Programmed death ligand 2 (anti-PD-L2), anti-CD137, anti-CD40, anti-OX40 antibodies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 119 (Actual)
Dates: Start 2011-09-23 (Actual); Primary Completion 2014-12-01 (Actual); Study Completion 2019-05-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (14):
- United States (12):
  - Ucsf Helen Diller Family Comprehensive Cancer Center, San Francisco, California
  - Yale University School Of Medicine, New Haven, Connecticut
  - H. Lee Moffitt Cancer Center, Tampa, Florida
  - University Of Chicago Medical Center, Chicago, Illinois
  - The Bunting-Blaustein Cancer Research Building, Baltimore, Maryland
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Dana Farber Cancer Inst, Boston, Massachusetts
  - Duke University Medical Center, Durham, North Carolina
  - Providence Portland Med Ctr, Portland, Oregon
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Upmc Cancer Pavilion, Pittsburgh, Pennsylvania
  - University Of Wisconsin Carbone Cancer Center, Madison, Wisconsin
- Local Institution, Villejuif, France
- Local Institution, Pamplona, Spain

REFERENCES:
- [Derived] Ross-Macdonald P, Walsh AM, Chasalow SD, Ammar R, Papillon-Cavanagh S, Szabo PM, Choueiri TK, Sznol M, Wind-Rotolo M. Molecular correlates of response to nivolumab at baseline and on treatment in patients with RCC. J Immunother Cancer. 2021 Mar;9(3):e001506. doi: 10.1136/jitc-2020-001506. PMID 33658305
- [Derived] Zhou Q, Qi Y, Wang Z, Zeng H, Zhang H, Liu Z, Huang Q, Xiong Y, Wang J, Chang Y, Bai Q, Xia Y, Wang Y, Liu L, Xu L, Dai B, Guo J, Zhu Y, Zhang W, Xu J. CCR5 blockade inflames antitumor immunity in BAP1-mutant clear cell renal cell carcinoma. J Immunother Cancer. 2020 Apr;8(1):e000228. doi: 10.1136/jitc-2019-000228. PMID 32371459
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/s/US/English/USenHome
- See also: Investigator Inquiry Form — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 119 participants were enrolled, 92 participants were randomized of whom 1 was randomized but not treated. 27 participants did not enter treatment period due to: Participant withdrawal n = 1, Death n = 1, No longer meets criteria n = 22, Other reasons n = 3
Groups:
- Nivolumab 0.3 mg/kg (Previously-treated); Nivolumab 2 mg/kg (Previously-treated); Nivolumab 10 mg/kg (Previously-treated): Nivolumab was administered as a 60 minute IV infusion to participants who were previously treated with at least one anti-angiogenic therapy. Participants were dosed every 3 weeks until discontinuation or the end of the study.
- Nivolumab 10 mg/kg (Treatment-naive): Nivolumab was administered as a 60 minute IV infusion to treatment-naive participants. Participants were dosed every 3 weeks until discontinuation or the end of the study.
Period: Overall Study
Arm/Group | Nivolumab 0.3 mg/kg (Previously-treated) | Nivolumab 2 mg/kg (Previously-treated) | Nivolumab 10 mg/kg (Previously-treated) | Nivolumab 10 mg/kg (Treatment-naive)
Started | 22 | 22 | 23 | 24
Completed (Completed = continuing in the treatment period) | 1 | 0 | 1 | 0
Not Completed | 21 | 22 | 22 | 24
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1
Not completed — Death | 0 | 2 | 0 | 0
Not completed — Study Drug Toxicity | 1 | 3 | 4 | 5
Not completed — SUBJ request to discontinue study TRT | 0 | 0 | 0 | 1
Not completed — Subject No Longer Meets Study Criteria | 0 | 2 | 0 | 1
Not completed — Adverse Event related to study drug | 1 | 0 | 0 | 1
Not completed — Disease Progression | 19 | 15 | 17 | 15
Not completed — Out of State/Unmet Criteria | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Nivolumab 0.3 mg/kg (Previously-treated) | Nivolumab 2 mg/kg (Previously-treated) | Nivolumab 10 mg/kg (Previously-treated) | Nivolumab 10 mg/kg (Treatment-naive) | Total
Number analyzed (Participants) | 22 | 22 | 23 | 24 | 91
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.0 (.41) | 60.8 (9.89) | 57.7 (10.98) | 61.8 (10.3) | 60.3 (10.13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 10 | 8 | 9 | 30
  Male | 19 | 12 | 15 | 15 | 61
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1 | 1 | 3
  Not Hispanic or Latino | 16 | 19 | 17 | 23 | 75
  Unknown or Not Reported | 5 | 3 | 5 | 0 | 13
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 1 | 0 | 0 | 2
  White | 20 | 21 | 21 | 24 | 86
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in Activated and Memory T Cells
Description: The objective of the study was to investigate the pharmacodynamic immunomodulatory activity of anti-PD-1 antibody in activated and memory T cells with metastatic clear-cell Renal Cell Carcinoma (RCC)
Time Frame: Baseline, Cycle 1 Day 1, Cycle 1 Day 2, Cycle 1 Day 8, Cycle 2 Day 8, Cycle 4 Day 1
Population: All participants in the biomarker data set with baseline measurement and at least one on treatment measurement were included in pharmacodynamic analyses.
Measure: Mean (95% Confidence Interval); unit: Percentage
Arm/Group | Nivolumab 0.3 mg/kg (Previously-treated) | Nivolumab 2 mg/kg (Previously-treated) | Nivolumab 10 mg/kg (Previously-treated) | Nivolumab 10 mg/kg (Treatment-naive)
Number analyzed (Participants) | 22 | 22 | 23 | 24
Percentage
  Cycle 1 Day 1 | NA [NA to NA] — Due to improper storage at the central laboratory resulting in poor cell viability, the peripheral blood mononuclear cell (PBMC) samples were unable to be tested for activated and memory T cells | NA [NA to NA] — Due to improper storage at the central laboratory resulting in poor cell viability, the peripheral blood mononuclear cell (PBMC) samples were unable to be tested for activated and memory T cells | NA [NA to NA] — Due to improper storage at the central laboratory resulting in poor cell viability, the peripheral blood mononuclear cell (PBMC) samples were unable to be tested for activated and memory T cells | NA [NA to NA] — Due to improper storage at the central laboratory resulting in poor cell viability, the peripheral blood mononuclear cell (PBMC) samples were unable to be tested for activated and memory T cells
  Cycle 1 Day 2 | NA [NA to NA] — Due to improper storage at the central laboratory resulting in poor cell viability, the peripheral blood mononuclear cell (PBMC) samples were unable to be tested for activated and memory T cells | NA [NA to NA] — Due to improper storage at the central laboratory resulting in poor cell viability, the peripheral blood mononuclear cell (PBMC) samples were unable to be tested for activated and memory T cells | NA [NA to NA] — Due to improper storage at the central laboratory resulting in poor cell viability, the peripheral blood mononuclear cell (PBMC) samples were unable to be tested for activated and memory T cells | NA [NA to NA] — Due to improper storage at the central laboratory resulting in poor cell viability, the peripheral blood mononuclear cell (PBMC) samples were unable to be tested for activated and memory T cells
  Cycle 1 Day 8 | NA [NA to NA] — Due to improper storage at the central laboratory resulting in poor cell viability, the peripheral blood mononuclear cell (PBMC) samples were unable to be tested for activated and memory T cells | NA [NA to NA] — Due to improper storage at the central laboratory resulting in poor cell viability, the peripheral blood mononuclear cell (PBMC) samples were unable to be tested for activated and memory T cells | NA [NA to NA] — Due to improper storage at the central laboratory resulting in poor cell viability, the peripheral blood mononuclear cell (PBMC) samples were unable to be tested for activated and memory T cells | NA [NA to NA] — Due to improper storage at the central laboratory resulting in poor cell viability, the peripheral blood mononuclear cell (PBMC) samples were unable to be tested for activated and memory T cells
  Cycle 2 Day 8 | NA [NA to NA] — Due to improper storage at the central laboratory resulting in poor cell viability, the peripheral blood mononuclear cell (PBMC) samples were unable to be tested for activated and memory T cells | NA [NA to NA] — Due to improper storage at the central laboratory resulting in poor cell viability, the peripheral blood mononuclear cell (PBMC) samples were unable to be tested for activated and memory T cells | NA [NA to NA] — Due to improper storage at the central laboratory resulting in poor cell viability, the peripheral blood mononuclear cell (PBMC) samples were unable to be tested for activated and memory T cells | NA [NA to NA] — Due to improper storage at the central laboratory resulting in poor cell viability, the peripheral blood mononuclear cell (PBMC) samples were unable to be tested for activated and memory T cells
  Cycle 4 Day 1 | NA [NA to NA] — Due to improper storage at the central laboratory resulting in poor cell viability, the peripheral blood mononuclear cell (PBMC) samples were unable to be tested for activated and memory T cells | NA [NA to NA] — Due to improper storage at the central laboratory resulting in poor cell viability, the peripheral blood mononuclear cell (PBMC) samples were unable to be tested for activated and memory T cells | NA [NA to NA] — Due to improper storage at the central laboratory resulting in poor cell viability, the peripheral blood mononuclear cell (PBMC) samples were unable to be tested for activated and memory T cells | NA [NA to NA] — Due to improper storage at the central laboratory resulting in poor cell viability, the peripheral blood mononuclear cell (PBMC) samples were unable to be tested for activated and memory T cells

2. Primary Outcome: Mean Serum Cytokines: CXCL9
Description: Objective is to investigate the pharmacodynamic immunomodulatory activity of serum chemokines (CXCL9, CXCL10)
Time Frame: Baseline, Cycle 1 Day 1 3 Hrs Post, Cycle 1 Day 1 7 Hr Post, Cycle 1 Day 2 24 Hr Post, Cycle 2 Day 1 0 Hr Pre, Cycle 2 Day 8 168 Hrs Post, Cycle 4 Day 1 O Hr Pre (~39 months)
Population: Biomarker evaluable population: All treated participants with at least one measurement for a specific marker were included in the data set for that marker.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Nivolumab 0.3 mg/kg (Previously-treated) | Nivolumab 2 mg/kg (Previously-treated) | Nivolumab 10 mg/kg (Previously-treated) | Nivolumab 10 mg/kg (Treatment-naive)
Number analyzed (Participants) | 22 | 22 | 23 | 24
pg/mL
  Cycle 1 Day 1, 3 HRSPOST: number analyzed (Participants) | 22 | 22 | 22 | 23
  Cycle 1 Day 1, 3 HRSPOST | 2859.1 (2481.44) | 2294.3 (1528.97) | 1906.6 (1744.09) | 2203.6 (1728.76)
  Cycle 1 Day 1, 7HRSPOST: number analyzed (Participants) | 21 | 21 | 23 | 22
  Cycle 1 Day 1, 7HRSPOST | 3287.7 (3617.32) | 2567.1 (1885.13) | 2546.1 (2421.00) | 2883.6 (2827.77)
  Cycle 1 Day 2, 24 HRSPOST: number analyzed (Participants) | 21 | 21 | 23 | 23
  Cycle 1 Day 2, 24 HRSPOST | 5447.3 (7006.73) | 4332.3 (3875.12) | 4216.4 (4715.61) | 3858.80 (2841.7)
  Cycle 2 Day 1, 0 HRSPRE: number analyzed (Participants) | 21 | 19 | 23 | 23
  Cycle 2 Day 1, 0 HRSPRE | 5192.6 (4447.78) | 7220.6 (9385.90) | 5398.8 (5428.64) | 5687.4 (6788.78)
  Cycle 2 Day 8, 168 HRSPOST: number analyzed (Participants) | 20 | 19 | 23 | 22
  Cycle 2 Day 8, 168 HRSPOST | 5271.5 (5196.91) | 4932.6 (4321.91) | 5751.3 (5900.87) | 5773.2 (6560.9)
  Cycle 4 Day 1, 0 HRSPRE: number analyzed (Participants) | 15 | 17 | 16 | 21
  Cycle 4 Day 1, 0 HRSPRE | 8519.4 (11444.72) | 5131.2 (4330.84) | 3523.6 (2678.32) | 5449.5 (4021.84)
  BASELINE: number analyzed (Participants) | 22 | 21 | 23 | 24
  BASELINE | 2681.6 (2135.89) | 2213.5 (1520.44) | 2065.3 (1805.25) | 2610.6 (2118.11)

3. Primary Outcome: Mean Serum Cytokines CXCL10 (IP10)
Description: Objective is to investigate the pharmacodynamic immunomodulatory activity of serum chemokines (CXCL9, CXCL10)
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Nivolumab 0.3 mg/kg (Previously-treated) | Nivolumab 2 mg/kg (Previously-treated) | Nivolumab 10 mg/kg (Previously-treated) | Nivolumab 10 mg/kg (Treatment-naive)
Number analyzed (Participants) | 22 | 22 | 23 | 24
pg/mL
  Cycle 1 Day 1, 3 HRSPOST: number analyzed (Participants) | 22 | 22 | 22 | 23
  Cycle 1 Day 1, 3 HRSPOST | 525.5 (335.10) | 523.4 (400.88) | 422.0 (264.54) | 450.7 (247.78)
  Cycle 1 Day 1, 7HRSPOST: number analyzed (Participants) | 21 | 21 | 23 | 22
  Cycle 1 Day 1, 7HRSPOST | 591.4 (360.30) | 727.7 (626.98) | 762.2 (896.22) | 531.4 (508.20)
  Cycle 1 Day 2, 24 HRSPOST: number analyzed (Participants) | 21 | 21 | 23 | 23
  Cycle 1 Day 2, 24 HRSPOST | 813.2 (547.71) | 758.8 (616.06) | 736.1 (787.53) | 700.5 (738.71)
  Cycle 2 Day 1, 0 HRSPRE: number analyzed (Participants) | 21 | 19 | 23 | 23
  Cycle 2 Day 1, 0 HRSPRE | 718.0 (471.22) | 835.9 (579.07) | 781.9 (753.41) | 679.4 (556.47)
  Cycle 2 Day 8, 168 HRSPOST: number analyzed (Participants) | 20 | 19 | 23 | 22
  Cycle 2 Day 8, 168 HRSPOST | 724.1 (470.03) | 677.6 (341.15) | 794.6 (882.64) | 770.6 (672.43)
  Cycle 4 Day 1, 0 HRSPRE: number analyzed (Participants) | 15 | 17 | 16 | 21
  Cycle 4 Day 1, 0 HRSPRE | 1272.8 (2075.49) | 678.7 (364.85) | 431.3 (133.78) | 794.8 (574.14)
  BASELINE: number analyzed (Participants) | 22 | 21 | 23 | 24
  BASELINE | 474.5 (236.75) | 483.0 (383.77) | 397.4 (223.89) | 767.9 (525.06)

4. Primary Outcome: Mean CD4 T Cell Infiltration
Description: The objective of the study was to investigate the pharmacodynamic immunomodulatory activity of anti-PD-1 antibody on circulating CD4 infiltrations in tumors in participants with metastatic clear-cell Renal Cell Carcinoma (RCC).
Time Frame: Cycle 2 Day 8 168 Hr post dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Number of CD4+ Cells
Arm/Group | Nivolumab 0.3 mg/kg (Previously-treated) | Nivolumab 2 mg/kg (Previously-treated) | Nivolumab 10 mg/kg (Previously-treated) | Nivolumab 10 mg/kg (Treatment-naive)
Number analyzed (Participants) | 18 | 20 | 14 | 16
Number of CD4+ Cells
  Baseline | 34.1 (78.40) | 10.4 (34.38) | 35.2 (77.44) | 53.2 (109.31)
  Cycle 2 Day 8, 168 HrsPost: number analyzed (Participants) | 13 | 13 | 13 | 12
  Cycle 2 Day 8, 168 HrsPost | 64.8 (77.22) | 28.2 (46.93) | 53.4 (97.98) | 107.4 (254.75)

5. Primary Outcome: Mean CD8 T Cell Infiltration
Description: The objective of the study was to investigate the pharmacodynamic immunomodulatory activity of anti-PD-1 antibody on circulating CD8 infiltrations in tumors in participants with metastatic clear-cell Renal Cell Carcinoma (RCC).
Time Frame: 168 hour post does Cycle 2 Day 8 in evaluable participates (First active dose of study medication to cycle two day eight post injection)
Population: Biomarker evaluable population: All treated participants at least one measurement for a specific marker were included in the data set for that marker.
Measure: Mean (Standard Deviation); unit: Number of CD8 cells
Arm/Group | Nivolumab 0.3 mg/kg (Previously-treated) | Nivolumab 2 mg/kg (Previously-treated) | Nivolumab 10 mg/kg (Previously-treated) | Nivolumab 10 mg/kg (Treatment-naive)
Number analyzed (Participants) | 18 | 20 | 14 | 16
Number of CD8 cells
  Baseline: number analyzed (Participants) | 18 | 19 | 14 | 16
  Baseline | 10.2 (13.77) | 7.8 (10.62) | 11.9 (14.31) | 14.4 (18.37)
  Cycle 2 Day 8, 169 HRSPOST: number analyzed (Participants) | 13 | 13 | 13 | 12
  Cycle 2 Day 8, 169 HRSPOST | 14.9 (13.85) | 18.9 (17.07) | 23.3 (23.49) | 16.3 (22.19)

6. Secondary Outcome: Best Overall Response in the BMS-936558 Arms
Description: Baseline and post-nivolumab treatment modulation of serum levels of interferon-gamma stimulated chemokines CXCL9 and CXCL10 (IP10) were assessed. The participant's best response designation over the study as a whole, recorded between the date of first study drug administration and the date of objectively documented progression per Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST 1.1) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR
Time Frame: Assessed at a minimum of every 3 weeks up to 70 days following discontinuation of study drug (up to approximately 39 months)
Population: All treated participants
Measure: Count of Participants; unit: Participants
Arm/Group | Nivolumab 0.3 mg/kg (Previously-treated) | Nivolumab 2 mg/kg (Previously-treated) | Nivolumab 10 mg/kg (Previously-treated) | Nivolumab 10 mg/kg (Treatment-naive)
Number analyzed (Participants) | 22 | 22 | 23 | 24
Participants
  Complete Response | 0 | 0 | 0 | 2
  Partial Response | 2 | 4 | 5 | 1
  Stable Disease | 8 | 10 | 11 | 13
  Progressive Disease | 9 | 5 | 6 | 7
  Unable To Determine | 2 | 3 | 0 | 0

7. Secondary Outcome: Progression Free Survival Rate in BMS-936558
Description: PFS is defined as the time from treatment arm assignment to the date of first documented disease progression. Participants who die without a reported prior progression will be considered to have progressed on the date of their death. Participants who did not progress or die will be censored on the date of their last tumor assessment. Participants who did not have any on study tumor assessments will be censored on the date they were assigned a treatment arm. PFS rate is the percentage of participants who did not have disease progression at particular time points (16 weeks, 24 weeks, 48 weeks)
Time Frame: Progression free survival rate will be assessed in each individual treatment arm by tumor assessments at 16, 24, and 48 weeks. From initial dose to end of study (assessed up to 39 months)
Population: All treated participants
Measure: Number (95% Confidence Interval); unit: percent
Arm/Group | Nivolumab 0.3 mg/kg (Previously-treated) | Nivolumab 2 mg/kg (Previously-treated) | Nivolumab 10 mg/kg (Previously-treated) | Nivolumab 10 mg/kg (Treatment-naive)
Number analyzed (Participants) | 22 | 22 | 23 | 24
percent
  16 weeks | 0.29 [0.12 to 0.48] | 0.49 [0.27 to 0.68] | 0.63 [0.39 to 0.79] | 0.55 [0.32 to 0.72]
  24 weeks | 0 [0 to 0] | 0.44 [0.23 to 0.63] | 0.58 [0.35 to 0.76] | 0.50 [0.28 to 0.68]
  48 weeks | 0 [0 to 0] | 0 [0 to 0] | 0.32 [0.13 to 0.52] | 0.39 [0.18 to 0.59]

8. Secondary Outcome: Objective Response Rate in BMS-936558
Description: The total number of subjects whose best overall response (BOR) is either a complete response (CR) or partial response (PR) divided by the total number of participants in the population of interest, and expressed as a percentage.
Time Frame: Up to 22 months after study start
Population: All treated participants
Measure: Number (95% Confidence Interval); unit: percent
Arm/Group | Nivolumab 0.3 mg/kg (Previously-treated) | Nivolumab 2 mg/kg (Previously-treated) | Nivolumab 10 mg/kg (Previously-treated) | Nivolumab 10 mg/kg (Treatment-naive)
Number analyzed (Participants) | 22 | 22 | 23 | 24
percent | 9.1 [1.1 to 29.2] | 18.2 [5.2 to 40.3] | 21.7 [7.5 to 43.7] | 12.5 [2.7 to 32.4]

9. Secondary Outcome: Duration of Objective Response for BMS-936558
Description: The duration of response is defined as the time when the measurement criteria are first met for PR or CR (whichever is reported first) until the date of documented disease progression or death. For subjects who neither progress nor die, the duration of response will be censored at the date of their last tumor assessment.
Time Frame: The time when the measurement criteria are first met for PR or CR (whichever is reported first) until the date of documented disease progression or death (assessed up to 39 months)
Population: All treated participants
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Nivolumab 0.3 mg/kg (Previously-treated) | Nivolumab 2 mg/kg (Previously-treated) | Nivolumab 10 mg/kg (Previously-treated) | Nivolumab 10 mg/kg (Treatment-naive)
Number analyzed (Participants) | 22 | 22 | 23 | 24
weeks | 30 [24.1 to 35.9] | NA [NA to NA] — NA=Not Reached due to a high percentage of ongoing responders | 48.1 [12.0 to NA] — NA=Not Reached due to a high percentage of ongoing responders | NA [NA to NA] — NA=Not Reached due to a high percentage of ongoing responders

10. Secondary Outcome: Duration of Stable Disease for BMS-936558 as Measured in Participants Whose Best Overall Response is Stable Disease as the Time From Baseline Until the Date of Documented Disease Progression or Death
Description: Duration of stable disease (SD) is defined in participants whose BOR is SD at the time from treatment arm assignment until the criteria for progression are met or death (whichever occurs first). Participants who die without a reported prior progression will be considered to have progressed on the date of their death. Participants who did not progress or die will be censored on the date of their last tumor assessment
Time Frame: The time from treatment arm assignment until the criteria for progression are met or death (whichever occurs first)(assessed up to 39 months)
Population: All treated participants
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Nivolumab 0.3 mg/kg (Previously-treated) | Nivolumab 2 mg/kg (Previously-treated) | Nivolumab 10 mg/kg (Previously-treated) | Nivolumab 10 mg/kg (Treatment-naive)
Number analyzed (Participants) | 22 | 22 | 23 | 24
weeks | 16.5 [11.6 to 36.3] | 31.4 [10.7 to NA] — Upper limit not reached | 41.3 [12.1 to 75.6] | 35.1 [12.3 to 53.4]

11. Secondary Outcome: Immunogenicity of BMS-936558 as Measured by the Detection of Human Antibodies Against BMS-936558
Description: Blood samples to evaluate the development of a positive anti-drug antibodies (ADA) response at the doses tested will be collected at time-points pre-dose, C4D1, C8D1 and during follow-up.
Time Frame: Pre-dose, Cycle 4 Day 1, Cycle 8 Day 1 and during follow-up.
Population: ADA-Positive Subject: A subject with at least one ADA-positive sample at any time after initiation of treatment.
  ADA-Negative Subject: A subject with no ADA-positive sample after the initiation of treatment
Measure: Number; unit: percentage
Arm/Group | Nivolumab 0.3 mg/kg (Previously-treated) | Nivolumab 2 mg/kg (Previously-treated) | Nivolumab 10 mg/kg (Previously-treated) | Nivolumab 10 mg/kg (Treatment-naive)
Number analyzed (Participants) | 17 | 19 | 22 | 21
percentage
  Anti-Drug Antibody (ADA) positive (%) | 11.8 | 15.8 | 13.6 | 0
  Anti-Drug Antibody (ADA) negative(%) | 88.2 | 84.2 | 86.4 | 100

ADVERSE EVENTS:
Time Frame: From first dose to within 100 days of last dose. (10/2011 - 01/2015). From First dose up to 100 days after last dose of study drug, assessed up to January 2017 (approximately 39 months)
Groups:
- BMS 0.3 mg/kg; BMS 2 mg/kg; BMS 10 mg/kg: Nivolumab was administered as a 60 minute IV infusion to participants who were previously treated with at least one anti-angiogenic therapy. Participants were dosed every 3 weeks until discontinuation or the end of the study.
- BMS 10 mg/Kg-N: Nivolumab was administered as a 60 minute IV infusion to treatment-naive participants. Participants were dosed every 3 weeks until discontinuation or the end of the study.
Arm/Group | BMS 0.3 mg/kg | BMS 2 mg/kg | BMS 10 mg/kg | BMS 10 mg/Kg-N
Serious Adverse Events (participants affected / at risk) | 13/22 | 11/22 | 12/23 | 13/24
Other Adverse Events (participants affected / at risk) | 22/22 | 22/22 | 23/23 | 24/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | BMS 0.3 mg/kg (N=22) | BMS 2 mg/kg (N=22) | BMS 10 mg/kg (N=23) | BMS 10 mg/Kg-N (N=24)
Atrial flutter (Cardiac disorders) | 0 | 0 | 1 | 0
Papilloedema (Eye disorders) | 0 | 0 | 0 | 1
Colitis (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Constipation (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Enteritis (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Small intestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Pain (General disorders) | 0 | 0 | 0 | 1
Pyrexia (General disorders) | 1 | 0 | 0 | 0
Sudden death (General disorders) | 0 | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 1
Viral upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Tendon rupture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 2 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 2 | 0
Blood bilirubin increased (Investigations) | 0 | 0 | 2 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Polyarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 4 | 1 | 3
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Metastases to testicle (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Central nervous system necrosis (Nervous system disorders) | 1 | 0 | 0 | 0
Cerebral haemorrhage (Nervous system disorders) | 0 | 0 | 0 | 1
Tremor (Nervous system disorders) | 0 | 1 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 1 | 2 | 0
Renal colic (Renal and urinary disorders) | 1 | 0 | 0 | 0
Renal failure (Renal and urinary disorders) | 1 | 0 | 0 | 0
Renal mass (Renal and urinary disorders) | 0 | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 1
Embolism (Vascular disorders) | 0 | 1 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Haematemesis (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Bile duct obstruction (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Sepsis (Infections and infestations) | 0 | 1 | 0 | 0
Septic shock (Infections and infestations) | 0 | 0 | 0 | 1
Thermal burn (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Amylase increased (Investigations) | 0 | 0 | 0 | 1
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 1 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Ataxia (Nervous system disorders) | 0 | 0 | 1 | 0
Facial nerve disorder (Nervous system disorders) | 0 | 0 | 1 | 0
Ischaemic stroke (Nervous system disorders) | 1 | 0 | 0 | 0
Paralysis (Nervous system disorders) | 0 | 0 | 0 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 0 | 1 | 0
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Thrombosis (Vascular disorders) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | BMS 0.3 mg/kg (N=22) | BMS 2 mg/kg (N=22) | BMS 10 mg/kg (N=23) | BMS 10 mg/Kg-N (N=24)
Anaemia (Blood and lymphatic system disorders) | 6 | 1 | 6 | 4
Hypothyroidism (Endocrine disorders) | 1 | 1 | 4 | 2
Eye pruritus (Eye disorders) | 0 | 1 | 0 | 2
Vision blurred (Eye disorders) | 0 | 0 | 0 | 2
Abdominal discomfort (Gastrointestinal disorders) | 0 | 1 | 0 | 2
Abdominal distension (Gastrointestinal disorders) | 1 | 2 | 2 | 0
Abdominal pain (Gastrointestinal disorders) | 6 | 3 | 3 | 5
Abdominal pain upper (Gastrointestinal disorders) | 3 | 1 | 2 | 1
Constipation (Gastrointestinal disorders) | 7 | 6 | 5 | 6
Diarrhoea (Gastrointestinal disorders) | 4 | 4 | 5 | 9
Dry mouth (Gastrointestinal disorders) | 1 | 2 | 1 | 5
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 3 | 0
Nausea (Gastrointestinal disorders) | 8 | 7 | 6 | 10
Vomiting (Gastrointestinal disorders) | 3 | 4 | 3 | 3
Asthenia (General disorders) | 2 | 2 | 4 | 2
Chest pain (General disorders) | 2 | 0 | 2 | 0
Chills (General disorders) | 2 | 3 | 3 | 4
Fatigue (General disorders) | 12 | 13 | 15 | 13
Mucosal inflammation (General disorders) | 0 | 0 | 1 | 3
Oedema peripheral (General disorders) | 4 | 2 | 7 | 3
Pain (General disorders) | 0 | 4 | 4 | 0
Pyrexia (General disorders) | 3 | 3 | 3 | 1
Cellulitis (Infections and infestations) | 1 | 2 | 0 | 0
Rash pustular (Infections and infestations) | 0 | 0 | 0 | 2
Rhinitis (Infections and infestations) | 3 | 0 | 0 | 1
Sinusitis (Infections and infestations) | 1 | 0 | 1 | 3
Upper respiratory tract infection (Infections and infestations) | 1 | 3 | 3 | 4
Urinary tract infection (Infections and infestations) | 3 | 1 | 0 | 0
Viral upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 2
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 2
Infusion related reaction (Injury, poisoning and procedural complications) | 1 | 1 | 4 | 4
Alanine aminotransferase increased (Investigations) | 2 | 0 | 2 | 2
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 3 | 2
Blood alkaline phosphatase increased (Investigations) | 1 | 3 | 2 | 0
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 2
Blood creatinine increased (Investigations) | 2 | 4 | 2 | 2
Weight decreased (Investigations) | 6 | 3 | 1 | 1
Decreased appetite (Metabolism and nutrition disorders) | 7 | 3 | 3 | 5
Dehydration (Metabolism and nutrition disorders) | 0 | 2 | 1 | 4
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 2 | 0 | 3
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 2 | 3 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 0 | 0 | 2
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 2 | 1 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 2 | 6 | 9
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 3 | 5 | 8
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 2
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 | 1 | 1 | 2
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2 | 2 | 2 | 4
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 3 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 2 | 2
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 3 | 2 | 3
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2 | 0 | 0
Dizziness (Nervous system disorders) | 3 | 2 | 3 | 4
Dysgeusia (Nervous system disorders) | 1 | 0 | 1 | 3
Headache (Nervous system disorders) | 4 | 5 | 3 | 1
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 2 | 2
Restless legs syndrome (Nervous system disorders) | 0 | 0 | 2 | 0
Depression (Psychiatric disorders) | 1 | 1 | 2 | 2
Insomnia (Psychiatric disorders) | 4 | 3 | 2 | 2
Mental status changes (Psychiatric disorders) | 0 | 2 | 0 | 0
Haematuria (Renal and urinary disorders) | 1 | 1 | 1 | 2
Urinary retention (Renal and urinary disorders) | 2 | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 7 | 8 | 4 | 5
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2 | 4
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 5 | 2 | 5
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 3 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 3
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 3 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 2
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 2
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 1 | 1
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 3
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 1 | 1 | 3
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 2 | 0 | 2
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 3 | 4 | 4 | 4
Rash (Skin and subcutaneous tissue disorders) | 5 | 2 | 2 | 2
Rash pruritic (Skin and subcutaneous tissue disorders) | 1 | 0 | 2 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 1
Hypertension (Vascular disorders) | 1 | 2 | 2 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.